CLINICAL TRIAL: NCT04808713
Title: RESILIENT - An Online Multidimensional Treatment to Promote Resilience After a Disaster: Randomized Controlled Trial Protocol
Acronym: RESILIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Geneviève Belleville, Full professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-030
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Post Traumatic Stress Disorder; Insomnia; Depression
Keywords: mental health; post-traumatic stress disorder; psychological distress; sleep
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Depression; Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment condition (Experimental)
  Interventions: Behavioral: Treatment
- Waitlist condition (No Intervention)

INTERVENTIONS:
Behavioral: Treatment — The treatment is a therapist-assisted self-help online cognitive-behaviour therapy focusing on post-traumatic stress, sleep and mood. It includes 12 sessions of evidence-based psychotherapeutic components, such as psychoeducation about PTSD, sleep and depression; prolonged exposure to avoided situations and memories; sleep management strategies (restriction of time in bed, stimulus control, sleep hygiene education); behavioural activation; relaxation and mindfulness exercises; problem-solving strategies; and cognitive restructuring. A small portion of material was unlocked each week, and access to one module was accessible after the completion of a previous one. Supervised graduate psychology students provided brief regular weekly contacts for 12 weeks by video chat or phone, according to the participant's preference. Access to the online material was unlimited in time.
  Arms: Treatment condition

SUMMARY:
Background. The wildfires on May 1, 2016 in Fort McMurray, Alberta (Canada), destroyed approximately 2,400 homes and buildings and led to massive displacement of approximately 88,000 people. Many individuals faced direct or potential threat to their life or health, or significant losses, and many months later, families were still living through ongoing adversity and uncertainty as they adapted to new or temporary homes, schools and workplaces. Alberta Health Services estimated in August 2016 that mental health staff in the city had received 20,000 referrals since May, compared to 1,200 referrals each year.

Objectives. The overarching aim of this project is to understand the needs of the Fort McMurray population in terms of mental health and to widely disseminate evidence-based tools to promote resilience. More specifically, we will assess the efficacy of an online self-help intervention targeting post-traumatic resilience on specific symptoms (post-traumatic stress disorder [PTSD], insomnia, depression).

Method. 1,510 phone surveys have been conducted in May-July 2017 to assess the prevalence of PTSD, insomnia and depression in the evacuees from the Fort McMurray wildfires (T0). After the survey, 697 participants expressed interest to participate in the longitudinal arm of the study, which will include four in-depth assessments with online questionnaires (T1 to T4) and a diagnostic interview (T1 only). A period of six months will separate all four times of assessment. Participants with post-traumatic stress symptoms (expected n = 150) will be randomised either to the treatment condition (n = 75) or to a waitlist control condition (n = 75) after completion of T2.

Data Analyses. Primary outcomes will be post-traumatic, depressive and insomnia symptom severity, measured with validated self-report questionnaires. Secondary outcomes will include cognitive, behavioural and social indicators, as well as general mental health and post-traumatic growth. Several probable moderators of treatment will be examined, including sociodemographic characteristics, level of exposure, and continuing stressors.

Foreseen Impacts. If found effective in reducing symptoms, the results of this study have the potential to impact positively the Fort McMurray community. Indeed, a direct and concrete deliverable of this research project will be to provide an extended (at least two years) and free access to the online intervention specifically tailored to this population's needs.

ELIGIBILITY:
Inclusion Criteria:

* Significant post-traumatic stress symptoms (PCL-5 ≥ 23) OR
* Some post-traumatic stress symptoms (PCL-5 ≥ 10) with at least mild depressive symptoms (PHQ-9 ≥ 5) and/or subclinical insomnia symptoms (ISI ≥ 8).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Post-Traumatic Stress Disorder | 6 months
  PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) - This self-reported questionnaire includes 20 items on a 5-point Likert scale (from 0 = Not at all to 4 = Extremely) evaluating posttraumatic symptoms in the past month. The total score range between 0 and 80 with higher scores indicating higher symptoms severity.
Depression | 6 months
  Patient Health Questionnaire Depression Scale (PHQ-9) - This self-reported questionnaire includes nine items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day). Total severity scores range from 0 to 27, with a higher score indicating a higher severity.
Insomnia (ISI) | 6 months
  Insomnia Severity Index (ISI) - This self-reported questionnaire includes seven items rated on a 5-point Likert scale (from 0 = No problem to 4 = Very severe problem) that evaluate sleep difficulties in the past two weeks. Total severity scores range from 0 to 28, with a higher score indicating a higher severity of insomnia.

SECONDARY OUTCOMES:
Daily Functioning | 6 months
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) - This self-reported questionnaire includes 36 items on a 5-point Likert scale (from 0 = No difficulty to 4 = Extreme difficulty or cannot do) evaluating functioning in the past month and covering 6 domains: Understanding and Communicating (6 items), Getting around (5 items), Self-care (4 items), Getting along with others (5 items), Life activities (8 items), and Participation in society (8 items).
Generalized Anxiety Disorder | 6 months
  Patient Health Questionnaire Generalized Anxiety Disorder Scale (GAD-7) - This self-reported questionnaire includes 7 items on a 4-point Likert scale (from 0 = Not at all to 3 = Nearly every day) evaluating anxiety symptoms in the past two weeks. The total score range between 0 and 21 with higher scores indicating higher symptoms severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Background] Belleville G, Ouellet MC, Morin CM. Post-Traumatic Stress among Evacuees from the 2016 Fort McMurray Wildfires: Exploration of Psychological and Sleep Symptoms Three Months after the Evacuation. Int J Environ Res Public Health. 2019 May 8;16(9):1604. doi: 10.3390/ijerph16091604. PMID 31071909
- [Derived] Belleville G, Ouellet MC, Bekes V, Lebel J, Morin CM, Bouchard S, Guay S, Bergeron N, Ghosh S, Campbell T, Macmaster FP. Efficacy of a Therapist-Assisted Self-Help Internet-Based Intervention Targeting PTSD, Depression, and Insomnia Symptoms After a Disaster: A Randomized Controlled Trial. Behav Ther. 2023 Mar;54(2):230-246. doi: 10.1016/j.beth.2022.08.004. Epub 2022 Aug 19. PMID 36858756